CLINICAL TRIAL: NCT05606107
Title: To Compare the Efficacy and Safety of Low-dose Glucocorticoids and Tofacitinib in Alleviating Moderate to High Disease Activity Rheumatoid Arthritis for 24 Weeks
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jiaxing Hospital of T.C.M (Unknown); Jinhua Municipal Central Hospital (Other); SAHZU.CHANGXING CAMPUS (Unknown); Zhuji People's hospital (Unknown); Shaoxing People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0159
Record Dates: First submitted 2022-11-01; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis, moderate disease activity, high disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Glucocorticoids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid group (Active Comparator)
  Interventions: Drug: Glucocorticoid
- Tofacitinib group (Experimental)
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib combined with other csDMARDs, but no glucocorticoids.
  Arms: Tofacitinib group
Drug: Glucocorticoid — Glucocorticoid
  Arms: Glucocorticoid group

SUMMARY:
Glucocorticoids are effective in the treatment of rheumatoid arthritis, but long-term use of glucocorticoids has many side effects. Tofacitinib is a new small-molecule drug targeting JAK, which has been found to act quickly. The aim of this clinical trial was to investigate the efficacy and safety of tofacitinib and low-dose glucocorticoids in inducing remission in patients with rheumatoid arthritis with moderate to high disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years;
2. met the 2010 ACR and EULAR diagnostic criteria for rheumatoid arthritis (RA), and was diagnosed as RA;
3. After more than 3 months of initial treatment or conventional DMARDs treatment, the disease was still in medium-high disease activity, and DAS28-CRP>3.2;
4. No birth plan during and within 3 months after the end of the study;
5. Voluntarily sign the informed consent form.

Exclusion Criteria:

1. Patients who are using or have used glucocorticoids, tofacitib and biological agents in the past 3 months;
2. At the time of screening, patients were in the acute phase of acute infection or chronic infection;
3. Laboratory test results: Hb<100g/L; White blood cell count <4.0×10^9/L; Platelets <100×10^9/L; Liver function (transaminase, bilirubin)> 2 times the upper limit of normal value; Renal function (SCr) > the upper limit of normal;
4. Active gastrointestinal disease: gastrointestinal bleeding or active gastrointestinal ulcer and acute gastric mucosal injury diagnosed by gastroenteroscopy in the past three months;
5. A history of severe cardiovascular, cerebrovascular, kidney and other important organs, blood and endocrine system lesions, malignant tumors and thrombosis;
6. suffering from serious, progressive and uncontrolled diseases of other important organs and systems;
7. mental disease patients;
8. Other conditions deemed unsuitable for trial participation by the investigator;
9. Pregnancy tests of women of childbearing age were positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DAS28-CRP | 24 weeks
  Disease activity

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Changxing Country People's Hospital, Changxing
  - Jiaxing Central Hospital, Jiaxing
  - Jinhua Central Hospital, Jinhua
  - Shaoxing Central Hospital, Shaoxing
  - Zhuji People's Hospital, Zhuji